CLINICAL TRIAL: NCT02474628
Title: Consistencies in Responses to Sodium Bicarbonate Supplementation: a Randomised, Repeated Measures, Counterbalanced and Double-blind Study
Brief Title: Consistencies in Responses to Sodium Bicarbonate?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: Sodium bicarbonate consistency
Record Dates: First submitted 2015-06-08; First posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Sports Nutritional Physiological Phenomena
Keywords: Physiological Phenomena
MeSH Terms: interventions — Sodium Bicarbonate; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 0.3 g∙kg-1body mass of calcium carbonate
  Interventions: Dietary Supplement: calcium carbonate
- Sodium bicarbonate (Experimental): 0.3 g∙kg-1body mass of sodium bicarbonate
  Interventions: Dietary Supplement: sodium bicarbonate

INTERVENTIONS:
Dietary Supplement: sodium bicarbonate
  Arms: Sodium bicarbonate
Dietary Supplement: calcium carbonate
  Arms: Placebo

SUMMARY:
Intervention studies do not account for high within-individual variation potentially compromising the magnitude of an effect. Repeat administration of a treatment allows quantification of individual responses and determination of the consistency of responses. The investigators aim to determine the consistency of metabolic and exercise responses following repeated administration of sodium bicarbonate (SB). Design and Methods: 15 physically active males will complete six cycling capacity tests at 110% of maximum power output (CCT110%) following ingestion of either 0.3 g∙kg-1Body Mass of SB (4 trials) or placebo (PL, 2 trials). Blood pH, bicarbonate, base excess and lactate will be determined at baseline, pre-exercise, post-exercise and 5-min post-exercise. Total work done (TWD) will be recorded as the exercise outcome.

ELIGIBILITY:
Inclusion Criteria:

* recreationally active males

Exclusion Criteria:

* use of dietary supplements in the past 6 months
* the presence of any musculoskeletal disorder
* the use of anabolic steroids

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
blood pH | 5 min after a physical exercise test

SECONDARY OUTCOMES:
blood bicarbonate | 5 min after a physical exercise test
blood lactate | 5 min after a physical exercise test
anaerobic exercise capacity | 4 hours after supplementation
  as assessed by cycling capacity tests at 110% of maximum power output

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Froio de Araujo Dias G, da Eira Silva V, de Salles Painelli V, Sale C, Giannini Artioli G, Gualano B, Saunders B. (In)Consistencies in Responses to Sodium Bicarbonate Supplementation: A Randomised, Repeated Measures, Counterbalanced and Double-Blind Study. PLoS One. 2015 Nov 17;10(11):e0143086. doi: 10.1371/journal.pone.0143086. eCollection 2015. PMID 26574755